CLINICAL TRIAL: NCT03172585
Title: Can High Frequency Transthoracic Sonography Play a Competition Role With High Resolution Computed Tomography in Assessment of Alveolar Intersitial Syndrome
Brief Title: Transthoracic Sonography Versus High Resolution Computed Tomography in Alveolar Intersitial Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mariam hany adeeb, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AIS
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Resolution computed tomography (Other): Patients will be included in the study when High resolution chest computed tomography without contrast enhancement is ordered by the primary physician. Before the High resolution chest computed tomography scan, a Trans thoracic ultrasonography will be performed.
  Interventions: Other: High resolution computed tomography; Other: trans thoracic ultrasonography

INTERVENTIONS:
Other: High resolution computed tomography — High resolution computed tomography of the chest is the gold standard imaging modality for most pulmonary diseases
Other: trans thoracic ultrasonography — Trans thoracic ultrasonograghy is used progressively for evaluation of pulmonary diseases . Its non invasive nature , relatively low price ,portability for bedside use, and high reproducible of results allows for incorporation of imaging findings with clinical data

SUMMARY:
High resolution computed tomography of the chest is the gold standard imaging modality for most pulmonary diseases. However, the associated high expenses, radiation exposure , and its limited possibility for bedside use are a limitation.

DETAILED DESCRIPTION:
High resolution computed tomography of the chest is the gold standard imaging modality for most pulmonary diseases. However, the associated high expenses, radiation exposure , and its limited possibility for bedside use are a limitation. Transthoracic ultrasonograghy is used progressively for evaluation of pulmonary diseases. Its non invasive nature , relatively low price ,portability for bedside use, and high reproducibility of results allows for incorporation of imaging findings with clinical data. Although Transthoracic ultrasonograghy is not an alternative to High resolution computed tomography,it can potentially provide useful supplemental information in certain specific situations ,such as for rapid bedside diagnostic assessment of dyspneic patients. B-line is a common and significant abnormal sign used for diagnostic appraisal by Transthoracic ultrasonograghy, but it cannot define the exact underlying pathologic feature on a lung ultrasound. When the lung parenchymal pathology reaches the lung surface ,certain characteristic changes of the pleural line can be detected by means of the good imaging made possible by high-resolution Transthoracic ultrasonograghy ,but the application and strength of pleural line abnormalities in the differential diagnosis of lung diseases has not been adequately explored . Existing literature on the illustration of the pleural line is scarce ,and the shape of pleural line has not been adequately investigated and described ,especially in comparison with Computed tomography findings. Most studies that have investigated pleural lines are confined to the sub population with interstitial lung diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with dyspnea due to interstitial fibrosis syndrome.
2. pulmonary edema due to any cause.

Exclusion Criteria:

1. Traumatic lesions
2. Pneumothorax
3. Subcutaneous emphysema
4. Massive pleural effusion with atelectasis, and

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
the number of patients diagnosed with pleural diseases by high resolution computed tomography | 30 minutes
  computed tomography on the chest

CONTACTS AND LOCATIONS:
Overall Officials: Manal Mohamed, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sartori S, Tombesi P. Emerging roles for transthoracic ultrasonography in pleuropulmonary pathology. World J Radiol. 2010 Feb 28;2(2):83-90. doi: 10.4329/wjr.v2.i2.83. PMID 21160921
- [Background] Frenz MB, Mee AS. Diagnostic radiation exposure and cancer risk. Gut. 2005 Jun;54(6):889-90. doi: 10.1136/gut.2005.066605. No abstract available. PMID 15888804
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Smargiassi A, Inchingolo R, Soldati G, Copetti R, Marchetti G, Zanforlin A, Giannuzzi R, Testa A, Nardini S, Valente S. The role of chest ultrasonography in the management of respiratory diseases: document II. Multidiscip Respir Med. 2013 Aug 9;8(1):55. doi: 10.1186/2049-6958-8-55. PMID 23937897
- [Background] Leech M, Bissett B, Kot M, Ntoumenopoulos G. Lung ultrasound for critical care physiotherapists: a narrative review. Physiother Res Int. 2015 Jun;20(2):69-76. doi: 10.1002/pri.1607. Epub 2014 Dec 29. PMID 25545613
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688